CLINICAL TRIAL: NCT01574781
Title: Development of Non-invasive Prenatal Diagnostic Test Based on Fetal DNA Isolated From Maternal Blood
Brief Title: Non-invasive Prenatal Diagnostic Validation Study
Acronym: NIPD
Status: Completed | Type: Observational
Sponsor: Natera, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GSN012
Record Dates: First submitted 2012-04-02; First posted 2012-04-10 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-06

CONDITIONS: Chromosome 13 Aneuploidy; Chromosome 18 Aneuploidy; Chromosome 21 Aneuploidy; Sex Chromosome Aberrations; Other Microdeletions
Keywords: Down syndrome; Trisomy 13; Trisomy 18; Microdeletions; Pregnancy; Non-invasive
MeSH Terms: conditions — Sex Chromosome Aberrations; Down Syndrome; Trisomy 13 Syndrome; Trisomy 18 Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal blood, paternal blood or cheek swab, paternal relative blood or cheek swab, fetal blood or tissue, POC tissue, and child cord blood or saliva.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Women with abnormal fetus: Women carrying fetus that is identified as chromosomally abnormal by CVS/Amniocentesis
  Interventions: Procedure: Blood draw
- Women experiencing miscarriage: Women identified as miscarrying, prior to any D&C or D&E procedure
  Interventions: Procedure: Blood draw
- Born children: The children born from women participating in other cohorts of the study.
  Interventions: Procedure: Cheek swab/Saliva Sampling
- Male relatives: The male partners (and presumed biological father of any fetuses/children) of women participating in other cohorts of the study or the biological father's brother and/or father.
  Interventions: Procedure: Blood draw; Procedure: Cheek swab/Saliva Sampling
- Non-pregnant women: Healthy women who are not pregnant
  Interventions: Procedure: Blood draw
- Pregnant women
  Interventions: Procedure: Blood draw

INTERVENTIONS:
Procedure: Blood draw — Blood is drawn at the appropriate time given their cohort inclusion.
  Other Names: Non-Invasive Prenatal Diagnosis; NIPD
  Groups: Male relatives; Non-pregnant women; Pregnant women; Women experiencing miscarriage; Women with abnormal fetus
Procedure: Cheek swab/Saliva Sampling — In lieu of blood draw, male relatives may donate cheek swab or saliva sample. Children born to participating women can donate cheek swab or saliva sample soon after birth.
  Other Names: Non-Invasive Prenatal Diagnosis; NIPD
  Groups: Born children; Male relatives

SUMMARY:
The primary purpose of this study is to collect maternal blood samples from pregnant women to develop a non-invasive prenatal diagnostic test based on fetal DNA isolated from maternal blood.

DETAILED DESCRIPTION:
The investigators will seek to enroll subjects to collect the following types of samples:

* Up to 2,000 maternal blood samples along with their corresponding paternal blood, buccal or saliva samples (1,000 required for final analysis).
* Up to 200 maternal blood samples from carrying a fetus with a confirmed chromosomal abnormality or genetic disorder, along with their corresponding paternal blood, buccal or saliva samples (50 required for final analysis). For women who opted for termination, a genetic sample of the fetus may also be collected.
* Up to 1,000 buccal or saliva samples from paternal grandfathers and/or the biological father's brothers.
* Up to 1,000 cord, buccal or saliva samples from the born children.
* Up to 40 blood samples (20 non-pregnant females and 20 males) from healthy volunteers (20 required for final analysis)
* Up to 400 blood samples from women undergoing D&C procedure following a miscarriage along with corresponding paternal blood (or buccal or saliva samples) (200 required for final analysis).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who volunteer to donate blood sample during the first -, second- and/or third trimester
* The biological father of the child (or the father's brother and/or father) has to be at least 18 years of age and consent to his blood, buccal, or saliva collection.
* Pregnant women whose fetus was diagnosed with a chromosomal abnormality or genetic disorder by either amniocentesis or chorionic villus sampling who volunteer to donate a blood sample.
* Pregnant women who volunteer to donate a blood sample after their spontaneous miscarriage prior to undergoing D&C procedure and who choose to utilize Natera's commercial products of conception molecular karyotyping service.
* Healthy volunteers (non-pregnant female and male) who volunteer to donate their blood sample.
* Umbilical cord blood or cheek swab/saliva samples from born children o Pregnant women who have participated in donating a blood sample during their pregnancy have the option to donate either an umbilical cord blood sample after child delivery, or a cheek swab or saliva sample from the born child using Natera's home kit.

Exclusion Criteria:

* Women carrying multiples

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy non-pregnant women, pregnant women, male relatives, women undergoing miscarriage, and children born to participating women
Sampling Method: Non-Probability Sample
Enrollment: 1781 (Actual)
Dates: Start 2011-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Fetal chromosome abnormality from a maternal plasma sample | From date of initial blood draw until the date of pregnancy end (miscarriage/termination) or time of birth, whichever came first, assessed up to 10 months
  Maternal plasma will be drawn at the time at which they present while pregnant as long as they are at least 6 weeks along. Additional samples (for confirmation of chromosome makeup) may also be drawn on that fetus when fetal sampling is possible (termination, miscarriage) or on the child at or shortly after birth.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Rabinowitz, PhD, Principal Investigator — Natera, Inc.
Locations (1):
- Natera, Inc, Redwood City, California, United States